CLINICAL TRIAL: NCT03839992
Title: The Measurement and Analysis of Maximal Expiratory Flow Volume Loops at Low Lung Volumes in Children With Cystic Fibrosis and Normal Routine Lung Function.
Brief Title: Detection of Unsuspected Small Airways Obstruction in Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Gelb, Arthur F., M.D. (Individual)
Collaborators: Miller Children's & Women's Hospital Long Beach (Other); Stony Brook University (Other); The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Other Study IDs: MHS #843-18
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cystic Fibrosis in Children
Keywords: abnormal FEF75; bronchiectasis; lung CT
MeSH Terms: conditions — Bronchiectasis | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: spirometry — measure spirometry and lung CT

SUMMARY:
Goal is to physiologically detect unsuspected small airways obstruction in children and adults with treated heterozygous and homozygous cystic fibrosis. Unsuspected refers to normal routine pre bronchodilator spirometry including normal FEV1(L), FVC (L). and FEV1/FVC%. This is a retrospective study.

DETAILED DESCRIPTION:
The current study is based on current investigators previously published patho-physiologic and lung CT studies in small airways intrinsic obstruction, emphysema, and asthma. Current investigators have demonstrated that despite the presence of normal routine spirometry including normal FEV1(L), FVC (L), and FEV1/FVC% that unsuspected small airways obstruction, and emphysema can be detected. This has been achieved by presence of isolated abnormal expiratory airflow limitation at low lung volumes on the maximal expiratory flow volume curves. This includes abnormal expiratory airflow at 75% and 80% expired lung volume. Current investigators believe investigators will be able to detect unsuspected small airways intrinsic obstruction, and peripheral airway bronchiectasis proven by lung CT, in patients with cystic fibrosis despite presence of pre bronchodilator normal routine spirometry.

ELIGIBILITY:
Inclusion Criteria:

Heterozygote or homozygote patients with cystic fibrosis with normal routine pre bronchodilator spirometry including normal FEV1(L), FVC(L) and FEV1/FVC%.

Exclusion Criteria:Heterozygote or homozygote patients with cystic fibrosis with ABNORMAL routine pre bronchodilator spirometry

-

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Review pulmonary function and radiologic studies in retrospective records of heterozygote or homozygote patients with cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Detection of Unsuspected Small Airway Obstruction in Cystic Fibrosis | 5 years
  Retrospective analysis of pre bronchodilator spirometry, and lung CT study to detect abnormal FEF75% in the presence of normal spirometry and FEF25-75. Detect isolated abnormal pre bronchodilator spirometry at 75%FVC

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Gelb, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Arthur F Gelb MD, Lakewood, California
  - Miller Children's Hospital and Long Beach Medical Center, Long Beach, California

IPD SHARING:
Plan to Share IPD: Yes
All individual published data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: when published
Access Criteria: published data

REFERENCES:
- [Result] Mead J. The lung's "quiet zone". N Engl J Med. 1970 Jun 4;282(23):1318-9. doi: 10.1056/NEJM197006042822311. No abstract available. PMID 5442364
- [Result] Gelb AF, Gold WM, Wright RR, Bruch HR, Nadel JA. Physiologic diagnosis of subclinical emphysema. Am Rev Respir Dis. 1973 Jan;107(1):50-63. doi: 10.1164/arrd.1973.107.1.50. No abstract available. PMID 4683321
- [Result] Gelb AF, Zamel N. Simplified diagnosis of small-airway obstruction. N Engl J Med. 1973 Feb 22;288(8):395-8. doi: 10.1056/NEJM197302222880805. No abstract available. PMID 4684043
- [Result] Hogg JC, Pare PD, Hackett TL. The Contribution of Small Airway Obstruction to the Pathogenesis of Chronic Obstructive Pulmonary Disease. Physiol Rev. 2017 Apr;97(2):529-552. doi: 10.1152/physrev.00025.2015. PMID 28151425
- [Result] Lukic KZ, Coates AL. Does the FEF25-75 or the FEF75 have any value in assessing lung disease in children with cystic fibrosis or asthma? Pediatr Pulmonol. 2015 Sep;50(9):863-8. doi: 10.1002/ppul.23234. Epub 2015 Jun 16. PMID 26079395
- [Derived] Masson VK, Nussbaum E, Gelb AF, Tashkin DP, Randhawa I, Nadel JA, Fireizen Y, De Celie-Germana JK, Madera D, Senanayake D. Isolated abnormal FEF75% detects unsuspected bronchiolar obstruction in CF children. Pediatr Res. 2023 Sep;94(3):1051-1056. doi: 10.1038/s41390-023-02532-2. Epub 2023 Mar 13. PMID 36914809